CLINICAL TRIAL: NCT00674791
Title: A Phase I Study of Cancer Peptides Plus GM-CSF and Adjuvant (Montanide ISA 51) Following Completion of Prescribed Chemotherapy or Trastuzumab for TXN2-3M0 or Metastatic Breast Cancer With No Evidence of Disease
Brief Title: Study of Cancer Peptides Vaccine Plus GM-CSF as Adjuvant Treatment for High Risk (TXN2-3M0) or Metastatic Breast Cancer With No Evidence of Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Immunotope (Industry)
Responsible Party: Ramila Philip, Ph.D., Immunotope, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000902
Record Dates: First submitted 2008-05-05; First posted 2008-05-08 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2011-03

CONDITIONS: Breast Cancer
Keywords: Immunotherapeutic vaccine; breast cancer; TxN2-3M0 breast cancer; metastatic breast cancer; immunotherapy; antigen; Histologically confirmed, TxN2-3M0 or metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: OCPM Immunotherapeutic Vaccine — Patients will receive 1 injection into each thigh at each of 6 visits: week 0, week 1, week 2, week 4, week 5, and week 6. The first 9 patients will receive a 100 microgram dose and the second 9 patients a 1 milligram dose of the peptide mixture.

SUMMARY:
This study will evaluate the safety and feasibility of administering a peptide vaccine consisting of twelve different tumor-rejection antigens to patients with high risk (TxN2-3M0) or metastatic breast cancer with no evidence of disease following their completion of systemic therapy. The vaccine is designed to elicit immune responses against twelve different pathways that are essential to tumor growth, survival and metastasis.

DETAILED DESCRIPTION:
The primary endpoint will be to determine the safety and feasibility of administering cancer peptides to patients with high risk (TxN2-3M0) or metastatic breast cancer with no evidence of disease following their completion of systemic therapy, with the secondary objectives of evaluating immune response disease relapse survival. Two cohorts of 9 patients each will be treated with different doses of the vaccine. They will receive the peptide vaccine subcutaneously on weeks 0,1,2,4,5, and 6 and then receive the immunizations every 1 month for 6 months or disease recurrence. Toxicity will be assessed at each dose level using CTCv3 toxicity criteria.

ELIGIBILITY:
Inclusion Criteria:

* HLA-A2 patients with histologically confirmed, TxN2-3M0 or metastatic breast cancer with no evidence of disease who have completed their adjuvant systemic chemotherapy or trastuzumab
* Subjects will not be treated until 4 or more weeks after any prior chemotherapy, radiation therapy or immunotherapy, but they may be receiving hormonal therapy

Exclusion Criteria:

* History of autoimmune disease
* Serious intercurrent chronic or acute illness
* Active hepatitis
* Serologic evidence for HIV, splenectomy
* Receiving steroid or immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability: Number of subjects with dose limiting toxicity after 3 immunizations. | Status post-3 immunizations

SECONDARY OUTCOMES:
Immunologic response: Number of subjects with tumor antigen specific immune response after 3 immunizations. | Status post-3 immunizations

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morse, M.D., Principal Investigator — Duke University Cancer Center; Kimberly Blackwell, M.D., Principal Investigator — Duke University Cancer Center; Ramila Philip, Ph.D. — Immunotope
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States